CLINICAL TRIAL: NCT03125083
Title: Role of Inflammation in Psychiatric Disorders in Patients With Cutaneous Lupus
Acronym: RIP-LC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Société Française de Cardiologie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHU-316; 2017-A00336-47 (Other: 2017-A00336-47)
Record Dates: First submitted 2017-04-13; First posted 2017-04-24 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2019-08

CONDITIONS: Skin Restricted Lupus; Psychiatric Disorders
Keywords: Skin restricted lupus; Psychiatric disorders; Inflammation; Kynurenine pathway
MeSH Terms: conditions — Mental Disorders; Inflammation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- skin-restricted lupus (SRL) patients (Experimental): Role of inflammation in psychiatric disorders in patients with cutaneous lupus
  Interventions: Biological: Biological dosage from plasma

INTERVENTIONS:
Biological: Biological dosage from plasma — The purpose of this study is to determine the role of inflammation in the high prevalence of psychiatric disorders in skin-restricted lupus (SRL) patients. SRL is an inflammatory disease. Inflammation can lead to a decrease in the synthesis of neurotransmitters via the activation of the IDO enzyme and to induce the synthesis of neurotoxic molecules (kynurenin pathway). This leads to the development of psychiatric disorders.

SUMMARY:
The purpose of this study is to determine the role of inflammation in the high prevalence of psychiatric disorders in skin-restricted lupus (SRL) patients. SRL is an inflammatory disease. Inflammation can lead to a decrease in the synthesis of neurotransmitters via the activation of the IDO enzyme and to induce the synthesis of neurotoxic molecules (kynurenin pathway). This leads to the development of psychiatric disorders.

Investigator therefore want to compare inflammation and neurotransmitter synthesis in SRL patients according to the presence or absence of psychiatric disorders.

Investigator expect a decrease in neurotransmitter synthesis and activation of the kynurenin pathway in patients with a psychiatric disorder.

DETAILED DESCRIPTION:
The purpose of this study is to determine the role of inflammation in the high prevalence of psychiatric disorders in skin-restricted lupus (SRL) patients. SRL is an inflammatory disease. Inflammation can lead to a decrease in the synthesis of neurotransmitters via the activation of the IDO enzyme and to induce the synthesis of neurotoxic molecules (kynurenin pathway). This leads to the development of psychiatric disorders.

Investigator therefore want to compare inflammation and neurotransmitter synthesis in SRL patients according to the presence or absence of psychiatric disorders.

Investigator expect a decrease in neurotransmitter synthesis and activation of the kynurenin pathway in patients with a psychiatric disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cutaneous lupus:

Chronic (or discoid) cutaneous lupus during activity:

Either the typical chronic lupus plaque (associated with erythema, hyperkeratosis, atrophy) sitting on the photoexposed areas of the face and / or on the scalp; The erythematous forms in sheets are excluded in order not to include patients who may be ambiguous in diagnosis with systemic lupus.

Either form "tumidus" of chronic lupus. Typical cutaneous histology of chronic cutaneous lupus (orthokeratosis hyperkeratosis with horny plugs, thickening of the basal membrane area (PAS staining), lymphocytic infiltrate predominantly peri-necular but possibly having lichenoid aspects with vacuolation of the epidermal basal layer and cytoids).

sub-acute erythematous form in the course of evolution, thus defined Lesions distributed on the body's photoexposed areas, erythematous, squamous leaving scarred scars, the intensity of which is clearly aggravated by exposure to light.

Diagnostic histology compatible with diagnosis (hyperketatose orthokeratosique, middle and / or higher dermal lymphocytic infiltrate).

Presence of anti-Ro serum antibodies.

- Age greater than or equal to 18 years

Exclusion Criteria:

* Uncertain diagnosis of lupus
* Systemic lupus
* Presence of anti-native DNA antibodies at a rate> 1/80
* Proteinuria greater than 0.5g / 24h (or more than 3+),
* Presence of more than 3 American College of Rheumatology (ACR) criteria for the diagnosis of systemic lupus
* Other inflammatory dermatological pathology
* Chronic inflammatory disease (other than lupus)
* Diabetes
* Surgery in the previous month
* Immunosuppressive therapy
* Pregnant and lactating women
* Abuse or dependence on all poisons (except tobacco and alcohol)
* Mental retardation
* Illiteracy or not sufficiently fluent in French
* Patients under legal protection

Patients with acute inflammatory (and / or infectious, and / or traumatic) illness or who have taken an anti-inflammatory (other than for cutaneous lupus), analgesic, antihistamine or aspirin therapy within 15 days prior to inclusion Participate in the study, but will be offered to shift the inclusion. They may be included 15 days after an inflammatory disease or discontinuation of such treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Difference in IDO activation and neurotransmitters synthesis inhibition between SRL patients with and without psychiatric disorders. | Blood samples at day 1 and plasma analyses at the end of the study (when all patients will be included, up to 15 months)
  comparison of plasma:
  * kynurenine / tryptophan and 3-hydroxykynurenine / kynurenine ratios for IDO activation
  * serotonin / tryptophan) et tyrosine / phenylalanine ratios for neurotransmitters synthesis inhibition between SRL patients with and without psychiatric disorders.

SECONDARY OUTCOMES:
Difference in kynurenine pathway activation between SRL patients with and without psychiatric disorders. | Blood samples at day 1 and plasma analyses at the end of the study (when all patients will be included, up to 15 months)
  comparison of plasma kynurenic acid / kynurenine and quinolinic acid / kynurenine ratios between SRL patients with and without psychiatric disorders.
Difference in cytokine concentration between SRL patients with and without psychiatric disorders | Blood samples at day 1 and plasma analyses at the end of the study (when all patients will be included, up to 15 months)
  comparison of plasma TNFα, IFNα, IFNγ, IL1, IL1ᵦ, IL2, IL6, IL4, IL8, IL10, IL17, IL18 and CRP between SRL patients with and without psychiatric disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle JALENQUES, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France